CLINICAL TRIAL: NCT04439292
Title: MATCH Treatment Subprotocol H: Phase II Study of Dabrafenib and Trametinib in Patients With Tumors With BRAF V600E or V600K Mutations (Excluding Melanoma, Thyroid Cancer, Colorectal Adenocarcinoma, and Non-Small Cell Lung Cancer)
Brief Title: Testing Trametinib and Dabrafenib as a Potential Targeted Treatment in Cancers With BRAF Genetic Changes (MATCH-Subprotocol H)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03273; NCI-2020-03273 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-H (Other: ECOG-ACRIN Cancer Research Group); EAY131-H (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (dabrafenib, trametinib) (Experimental): Patients receive dabrafenib mesylate PO BID and trametinib dimethyl sulfoxide PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dabrafenib Mesylate; Drug: Trametinib Dimethyl Sulfoxide

INTERVENTIONS:
Drug: Dabrafenib Mesylate — Given PO
  Other Names: Dabrafenib Methanesulfonate; GSK2118436 Methane Sulfonate Salt; GSK2118436B; Tafinlar
Drug: Trametinib Dimethyl Sulfoxide — Given PO
  Other Names: Mekinist; Meqsel; Spexotras

SUMMARY:
This phase II MATCH treatment trial identifies the effects of trametinib and dabrafenib in patients whose cancer has genetic changes called BRAF V600 mutations. Dabrafenib may stop the growth of cancer by blocking BRAF proteins which may be needed for cell growth. Trametinib may stop the growth of cancer cells by blocking MEK proteins which, in addition to BRAF proteins, may also be needed for cell growth. Researchers hope to learn if giving trametinib with dabrafenib will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive dabrafenib mesylate orally (PO) twice daily (BID) and trametinib dimethyl sulfoxide PO once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have a BRAF V600E or, V600K, V600R or V600D mutation, or another aberration, as identified via the MATCH Master Protocol
* Prothrombin time (PT)/International normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.3 x institutional ULN; subjects receiving anticoagulation treatment may be allowed to participate with INR established within the therapeutic range prior to registration to treatment
* Patients must have an ECHO or a nuclear study (multigated aquisition scan [MUGA] or First Pass) within 4 weeks prior to registration to treatment and must not have a left ventricular ejection fraction (LVEF) < the institutional lower limit of normal (LLN). If the LLN is not defined at a site, the LVEF must be > 50% for the patient to be eligible
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have NONE of the following cardiac criteria:

  * Clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
* Patients who previously received monoclonal antibody therapy (eg. ipilimumab and others) must have stopped the prior therapy for 8 or more weeks before starting on trametinib and dabrafenib

Exclusion Criteria:

* Patients with a diagnosis of metastatic melanoma from a cutaneous, acral, mucosal, or unknown primary site are excluded
* Patients with a diagnosis of papillary thyroid cancer are excluded
* Patients with a diagnosis of colorectal adenocarcinoma are excluded
* Patients with a diagnosis of non-small cell lung cancer are excluded
* Patients with a history of interstitial lung disease or pneumonitis are excluded
* Patients must not have known hypersensitivity to dabrafenib and trametinib or compounds of similar chemical or biologic composition or to dimethyl sulfoxide (DMSO)
* Patients must not have a history or current evidence/risk of retinal vein occlusion (RVO). An eye exam is required at baseline
* Patients who previously received MEK inhibitors (including, but not limited to, trametinib, binimetinib, cobimetinib, selumetinib, RO4987655 (CH4987655), GDC-0623 and pimasertib) will be excluded
* Patients who previously received BRAF inhibitors (including, but not limited to, dabrafenib (Tafinlar), vemurafenib (PLX-4720) (Zelboraf), RAF265, LGX818 (encorafenib), RO5212054 (PLX3603), ARQ 736, XL281 (BMS-908662), CEP-32496, and the BRAF/MEK dual inhibitor (RO5126766) will be excluded
* Patients with prior exposure to dabrafenib or trametinib on another treatment subprotocol of the MATCH trial are excluded
* Current use of a prohibited medication. Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A or CYP2C8 are ineligible. Current use of, or intended ongoing treatment with: herbal remedies (e.g., St. John's wort), or strong inhibitors or inducers of P-glycoprotein (Pgp) or breast cancer resistance protein 1 (Bcrp1) should also be excluded
* Patients with a history of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection are excluded. An exception will be patients with cleared HBV and HCV infection which will be allowed on study
* Patients with history of RAS mutation-positive tumors are not eligible regardless of interval from the current study

  * NOTE: Prospective RAS testing is not required. However, if the results of previous RAS testing are known, they must be used in assessing eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2015-08-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
  ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among eligible and treated patients. Objective response rate is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. For each treatment arm, 90% two-sided binomial exact confidence interval will be calculated for ORR.

SECONDARY OUTCOMES:
Overall survival (OS) | Assessed every 3 months for =< 2 years and every 6 months for year 3
  OS is defined as time from treatment start date to date of death from any cause. Patients alive at the time of analysis are censored at last contact date. OS will be evaluated specifically for each drug (or step) using the Kaplan-Meier method.
Progression free survival (PFS) | Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
  PFS is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. PFS will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Erin R Macrae, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Salama AKS, Wang V, Macrae ER, Park JI, Chen HX, Gray RJ, McShane LM, Rubinstein LV, Patton D, Williams PM, Hamilton SR, Armstrong DK, Tricoli JV, Conley BA, Arteaga CL, Harris LN, O'Dwyer PJ, Chen AP, Flaherty KT. Phase II Study of Dabrafenib and Trametinib in Patients With Tumors With BRAFV600E Mutations: Updated Results From NCI-MATCH ECOG-ACRIN Trial (EAY131) Subprotocol H. JCO Precis Oncol. 2026 Jan;10:e2500338. doi: 10.1200/PO-25-00338. Epub 2026 Jan 14. PMID 41533998

DOCUMENTS (1):
  • Study Protocol (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT04439292/Prot_001.pdf